CLINICAL TRIAL: NCT06480448
Title: Effects of Treadmill Training on Cardio Respiratory Endurance and Constipation in Children With Cerebral Palsy
Brief Title: Treadmill Training Effects on Cardiorespiratory Endurance and Constipation in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RIPHAH/FR&AHS/letter-01826
Record Dates: First submitted 2024-04-29; First posted 2024-06-28 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Cardiopulmonary
Keywords: motor function

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional physical therapy (Experimental): This group will only getting conventional therapy which include core stability training, strength training, gait training through Parallel bar etc.
  Interventions: Other: Traditional physical herapy
- Treadmill training (Active Comparator): This group will getting treadmill training will be started along with conventional therapy group. Training protocol will be standardized and follow FITT protocol for 12 weeks.
  Interventions: Other: Treadmill training

INTERVENTIONS:
Other: Traditional physical herapy — core stability, strengthening exercises, stationary bicycle training and sustained strechinng exercises.
  Arms: Traditional physical therapy
Other: Treadmill training — Treadmill training for 20 minutes three time a week.
  Arms: Treadmill training

SUMMARY:
This study examines the impact of treadmill training on cardiorespiratory endurance and constipation in children with cerebral palsy (CP). Treadmill training is evaluated for its potential to improve cardiovascular fitness and alleviate constipation through its rhythmic movements. The findings shed light on the broader health benefits of treadmill interventions beyond motor function improvement in children with CP

DETAILED DESCRIPTION:
This research investigates the effects of treadmill training on two distinct yet interconnected aspects of health in children with cerebral palsy (CP): cardiorespiratory endurance and constipation.

The research employs a longitudinal design, with participants undergoing a structured treadmill training program tailored to their individual needs and abilities. Outcome measures include objective assessments of cardiorespiratory fitness (e.g., exercise stress tests, spirometry) and subjective evaluations of constipation symptoms (e.g., bowel diaries, symptom questionnaires). Additionally, the study examines potential correlations between improvements in cardiorespiratory endurance and changes in constipation severity, exploring the interplay between physical fitness and gastrointestinal function in children with CP.

By investigating the effects of treadmill training on both cardiorespiratory endurance and constipation, this research aims to provide a comprehensive understanding of the broader health benefits associated with exercise interventions in children with cerebral palsy. The findings may inform the development of integrated rehabilitation programs that address multiple aspects of health and well-being in this population, ultimately improving overall quality of life and functional outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age 4 to 12 years.
* Children having 1, or 2 on GMFCM.
* Children with spastic diplegic cerebral palsy.
* Children with well cognitive behavior.
* Children having 1 to 2 level on constipation assessment scale.
* Defecation frequency less than 3 time a week.

Exclusion Criteria:

* Misdiagnosed or not conform to Cerebral palsy.
* Children should be medically stable uncontrolled seizures.
* The children with mental retardation or other neurological disorders.
* Children with taking medication like muscle relaxant or laxative

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2024-04-28 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Constipation Assessment Scale (CAS) | Baseline - 12th Week
  One commonly used tool for assessing constipation in children is the "Rome IV Criteria," which is part of the Rome IV diagnostic criteria for functional gastrointestinal disorders. These criteria provide a standardized framework for diagnosing constipation based on specific symptoms and duration requirements
6-mintues walk test | Baseline - 12th Week
  The 6-Minute Walk Test (6MWT) is a standardized assessment used to measure a person's functional exercise capacity and endurance. During the test, individuals are instructed to walk as far as they can within a six-minute period along a flat, straight course. The test is typically conducted in a corridor or along a marked pathway, and the distance covered is recorded at the end of the test.
  Before the test begins, participants receive instructions on the procedure and are given the opportunity to ask questions. Baseline measurements such as heart rate, blood pressure, and oxygen saturation may be taken. Participants are encouraged to walk at a self-selected pace, and they are allowed to rest if needed during the test. However, the timer continues to run during rest periods.
Heart Rate | Baseline - 12th Week
  The number of pulses over a minute is the standard heart rate measurement. This can also be calculated by doubling the number of pulses felt over 30 seconds.
VO2 Max | Baseline - 12th Week
  VO2 max, or maximal oxygen consumption, refers to the maximum amount of oxygen that an individual can utilize during intense or maximal exercise. This measurement is generally considered the best indicator of cardiovascular fitness and aerobic endurance.
Respiratory Rate | Baseline - 12th Week

CONTACTS AND LOCATIONS:
Overall Officials: Waqar Ahmed Awan, PhD, Principal Investigator — Riphah International University
Locations (1):
- Rehman Medical Institute, Peshawar, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No